CLINICAL TRIAL: NCT01900275
Title: Urinary Heparanase Activity as a Predictor of Acute Kidney Injury in Critically Ill Adults
Status: Completed | Type: Observational
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Eric Schmidt, Assistant Professor of Medicine, Denver Health and Hospital Authority
Other Study IDs: COMIRB 13-0425; UL1TR000154 (NIH)
Record Dates: First submitted 2013-07-12; First posted 2013-07-16 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Sepsis; Trauma; Shock; Acute Kidney Injury
Keywords: Sepsis; Trauma; Shock; Acute kidney injury; Heparanase
MeSH Terms: conditions — Sepsis; Wounds and Injuries; Shock; Acute Kidney Injury | interventions — Urine Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine will be collected, centrifuged, and frozen
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic shock or major trauma: Patients admitted within 24 hours to ICU for septic shock or major trauma (ISS > 15). Septic shock is defined by sepsis with hypotension requiring >4 hours of vasopressor support over previous 24 hours.
  Interventions: Other: Urine collection

INTERVENTIONS:
Other: Urine collection — Collection of 5 ml urine from urinary collection device (e.g. foley catheter).

SUMMARY:
Across the world, the most common cause of dying in the ICU is a disease called "sepsis". Sepsis is a disease in which the body's protective response to infection becomes too intense, unnecessarily damaging important organs in the body. Kidney damage during sepsis is particularly bad, as a person's chance of survival drops significantly when he or she develops kidney failure. This study plans to learn more about how to detect (and thus prevent) kidney failure early in sepsis. The current tests doctors use only detect kidney failure once it's already happened. We must therefore find better ways of detecting kidney failure earlier, when there is still a chance to protect the kidneys.

In this study, patients will provide a one-time sample of urine. We will check this urine for signs of a protein called "heparanase", which we believe is important in early kidney failure. We will then see if high heparanase activity in urine predicts the risk of developing kidney failure. We will compare results from patients with sepsis with results from patients with trauma, allowing us to determine if heparanase is only important in sepsis kidney failure.

ELIGIBILITY:
Inclusion Criteria:

1. Septic shock or major trauma. Septic shock will be defined by standard criteria including (a) the presence of the systemic inflammatory response syndrome (SIRS), (b) evidence of infection, and (c) treatment with vasopressor medications for > 4 hours despite > 30 ml/kg intravenous crystalloid resuscitation. As a critically-ill comparator group, we will also enroll adult patients admitted (within 24 hours prior to screening) to the Denver Health Surgical ICU with major trauma, as defined by an Injury Severity Score of > 15.

Exclusion Criteria:

Exclusion criteria include anuria, prisoners, absence of a routinely-inserted urine collection device, or gross hematuria. Additionally, patients with known genitourinary malignancy will be excluded, given that cancers are known to overexpress heparanase. Additional exclusion criteria include age < 18 years, and pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adults admitted to the Denver Health MICU or SICU for either (a) septic shock or (b) major trauma.
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury | 72 hours
  Acute kidney injury will be determined using RIFLE criteria, based upon change in serum creatinine or urine output.

CONTACTS AND LOCATIONS:
Overall Officials: Eric P Schmidt, MD, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States

REFERENCES:
- [Derived] Schmidt EP, Overdier KH, Sun X, Lin L, Liu X, Yang Y, Ammons LA, Hiller TD, Suflita MA, Yu Y, Chen Y, Zhang F, Cothren Burlew C, Edelstein CL, Douglas IS, Linhardt RJ. Urinary Glycosaminoglycans Predict Outcomes in Septic Shock and Acute Respiratory Distress Syndrome. Am J Respir Crit Care Med. 2016 Aug 15;194(4):439-49. doi: 10.1164/rccm.201511-2281OC. PMID 26926297